CLINICAL TRIAL: NCT04152772
Title: Effect of tDCS Timing on Safety Memory in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mascha Frank, Associate Professor (Research), Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1346426-5; P20GM130452 (NIH)
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: PTSD
Keywords: safety memory; PTSD; tDCS; ventromedial prefrontal cortex; fear conditioning; context processing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Individuals deemed eligible for the study will be randomized to 1) receiving active tDCS during extinction learning; sham during extinction consolidation, 2) receiving sham during extinction learning; active tDCS during extinction consolidation, 3) receiving sham during extinction learning; sham during extinction consolidation. (Anticipated enrollment: 90 participants).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS during extinction learning followed by sham tDCS during consolidation (Active Comparator): Active tDCS will be applied during the extinction learning phase followed by sham tDCS during the consolidation phase.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS during extinction learning followed by active tDCS during consolidation (Active Comparator): Sham tDCS will be applied during the extinction learning phase followed by active tDCS during the consolidation phase.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS during extinction learning followed by sham tDCS during consolidation (Sham Comparator): Sham tDCS will be applied during the extinction learning phase followed by sham tDCS during the consolidation phase.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Active tDCS will consist of 15 minutes of 2 mA intensity once, either applied during or after extinction learning.

SUMMARY:
The primary purpose of this study is to investigate the effects of tDCS timing on extinction memory in PTSD. A total of 90 participants will be randomized equally across one of three groups:

1. One group receiving active stimulation during extinction followed by sham stimulation during consolidation
2. One group receiving sham stimulation during extinction followed by active stimulation during consolidation
3. One group receiving sham stimulation both during extinction and consolidation

This study also includes an online sub-study (Aim 2) focused on contextual processing along the PTSD spectrum. The online study tests if there is an association between threat and non-threat learning in contextual and non-contextual situations. A maximum of 500 participants will be recruited using an online, panel-based platform.

DETAILED DESCRIPTION:
This is a three-arm study composed of four to five visits over an approximate period of three weeks. Up to ninety participants are exposed to a fear conditioning, extinction, and extinction memory paradigm at three separate study visits (day 3-5); one of these study visits will include active or sham transcranial direct current stimulation (tDCS) for a period of 15 minutes. Skin conductance reactivity during extinction memory (day 5) is the primary outcome. Additional study procedures include a screening period (day 1) and two optional MRI scans, one done on study day 2 and one done on study day 5. As the completion of MRI scans are an optional study component, MRI-related data is not reported here.

SUB-STUDY: The objective of this sub-study is to test performance differences between contextual and non-contextual processing in individuals across the PTSD spectrum using an online, panel-based platform. Following a within-subjects study design, up to 500 adult participants, 18-89 years, will be asked to complete experimental tasks that assess contextual (configural) and non-contextual (elemental) threat and non-threat learning. They will also provide demographic information (age, sex, ethnicity) and complete questionnaires assessing self-reported PTSD, anxiety, and depression severity. As this sub-study does not reflect a randomized clinical trial (no groups, no randomization, no intervention), no further information is reported here.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of PTSD, assessed by the Structured Clinical Interview of DSM-5 (SCID);
2. aged 18-70;
3. ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent;
4. Stable psychiatric medication use or treatment for at least 6 weeks.

Exclusion Criteria:

1. Lifetime history of psychotic or bipolar disorder;
2. Current moderate or severe substance use disorder; if mild, not under the influence at time of study participation;
3. Acute suicidal or homicidal ideation as detected on screening instruments or in the investigator team's opinion, is likely to attempt suicide within 6 months;
4. current (or past) significant neurological disorder, injury, or other intracranial pathology including severe traumatic brain injury or lifetime history of a) seizure disorder b) primary or secondary CNS tumors c) stroke or d) cerebral aneurysm;
5. lifetime history of moderate or, current unstable medical conditions;
6. Any problems that would interfere with study participation, including MRI- or tDCS-related contraindications (e.g., implanted metallic devices/substances, metallic tattoos, pregnancy, claustrophobia, holes in the skull, skin abnormalities under stimulation sites), or indication of colorblindness, or presence of any other condition or circumstance that, in the opinion of the investigator team, has the potential to prevent study completion and/or inability to schedule visit days within the allotted time, and/or to have a confounding effect on outcome assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, PhD, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faucher CR, Doherty RA, Philip NS, Harle ASM, Cole JJE, Van't Wout-Frank M. Is there a neuroscience-based, mechanistic rationale for transcranial direct current stimulation as an adjunct treatment for posttraumatic stress disorder? Behav Neurosci. 2021 Dec;135(6):702-713. doi: 10.1037/bne0000487. Epub 2021 Aug 2. PMID 34338547

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Then Sham Transcranial Direct Current Stimulation: Participants received 2mA transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by sham tDCS for the same duration
- Sham Then Active Transcranial Direct Current Stimulation: Participants received sham transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by active, 2mA tDCS
- Sham Then Sham Transcranial Direct Current Stimulation: Participants received sham transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by sham tDCS
Period: Overall Study
Arm/Group | Active Then Sham Transcranial Direct Current Stimulation | Sham Then Active Transcranial Direct Current Stimulation | Sham Then Sham Transcranial Direct Current Stimulation
Started | 19 | 20 | 23
Completed | 19 | 20 | 22
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Then Sham Transcranial Direct Current Stimulation | Sham Then Active Transcranial Direct Current Stimulation | Sham Then Sham Transcranial Direct Current Stimulation | Total
Number analyzed (Participants) | 19 | 20 | 23 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant did not disclose their age
  years
    number analyzed (Participants) | 19 | 19 | 23 | 61
    (all) | 45.2 (14.7) | 46.9 (15.5) | 43.7 (16.6) | 45.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 21 | 49
  Male | 4 | 7 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 19 | 20 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 1 | 0 | 0 | 1
  White | 17 | 19 | 18 | 54
  More than one race | 0 | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Posttraumatic Stress Disorder (PTSD) Checklist for DSM-5 [Mean (Standard Deviation); unit: Average score on the PCL-5] — Self-report PTSD symptom severity as measured with the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). Scores range from 0 to 80, with higher scores indicating greater symptom severity. A score of 31 or higher suggests a probable diagnosis of PTSD
  Average score on the PCL-5 | 48.00 (12.34) | 44.80 (14.48) | 41.98 (15.52) | 44.73 (14.26)

OUTCOME MEASURES:

1. Primary Outcome: Skin Conductance Responses
Description: Main protocol: Threat reactivity as quantified by skin conductance responses to a conditioned and subsequently extinguished stimulus versus a never conditioned stimulus.
Time Frame: Study visit day 4: during administration of fear extinction memory.
Measure: Mean (Standard Error); unit: Skin conductance in microsiemens
Groups:
- Active tDCS During Extinction Learning Followed by Sham tDCS During Consolidation: Participants received 2mA transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by sham tDCS for the same duration
- Sham tDCS During Extinction Followed by Active tDCS During Consolidation: Participants received sham transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by active, 2mA tDCS
- Sham tDCS During Extinction Followed by Sham tDCS During Consolidation: Participants received sham transcranial direct current stimulation (tDCS) during extinction learning of conditioned threat, followed by sham tDCS
Arm/Group | Active tDCS During Extinction Learning Followed by Sham tDCS During Consolidation | Sham tDCS During Extinction Followed by Active tDCS During Consolidation | Sham tDCS During Extinction Followed by Sham tDCS During Consolidation
Number analyzed (Participants) | 19 | 19 | 21
Skin conductance in microsiemens | 0.075 (0.025) | 0.088 (0.026) | 0.057 (0.025)
Statistical Analysis 1: Comparison: Active tDCS During Extinction Learning Followed by Sham tDCS During Consolidation vs Sham tDCS During Extinction Followed by Active tDCS During Consolidation vs Sham tDCS During Extinction Followed by Sham tDCS During Consolidation; Comparison of groups (3) on skin conductance reactivity to the previously extinguished stimulus versus never conditioned stimulus during extinction recall; Test type: Superiority; p = 0.02, Mixed Models Analysis — Significant Group (3 levels) by Stimulus (CS- vs CS+ extinguished) interaction. A priori threshold for statistical significance was set at p<0.05

ADVERSE EVENTS:
Time Frame: One day, following active tDCS or sham stimulation
Description: A transcranial direct current stimulation side effects questionnaire was used following active tDCS or sham stimulation.
Groups:
- Group 1: Active tDCS During Extinction Learning and Sham tDCS During Consolidation: In group 1 active tDCS was applied during the extinction learning phase followed by sham tDCS during the consolidation phase.
  Transcranial direct current stimulation included 15 minutes of 2 mA intensity.
- Group 2: Sham tDCS During Extinction Learning and Active tDCS During Consolidation: In group 2 sham tDCS was applied during the extinction learning phase followed by active tDCS during the consolidation phase.
  Transcranial direct current stimulation included 15 minutes of 2 mA intensity.
- Group 3: Sham tDCS During Extinction Learning and Sham tDCS During Consolidation: In group 3 sham tDCS was applied during the extinction learning phase followed by sham tDCS during the consolidation phase.
  No transcranial direct current stimulation was applied.
Arm/Group | Group 1: Active tDCS During Extinction Learning and Sham tDCS During Consolidation | Group 2: Sham tDCS During Extinction Learning and Active tDCS During Consolidation | Group 3: Sham tDCS During Extinction Learning and Sham tDCS During Consolidation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 16/19 | 18/20 | 19/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Active tDCS During Extinction Learning and Sham tDCS During Consolidation (N=19) | Group 2: Sham tDCS During Extinction Learning and Active tDCS During Consolidation (N=20) | Group 3: Sham tDCS During Extinction Learning and Sham tDCS During Consolidation (N=23)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Neck or scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ringing or buzzing in ears (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Acute mood change (Psychiatric disorders) | 3 (3) | 2 (2) | 7 (7)
Difficulty concentrating (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Feeling sleepy or drowsy (Nervous system disorders) | 9 (9) | 12 (12) | 9 (9)
Experience of flickering lights (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1)
Feeling dizzy or lightheaded (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Feeling nauseous (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Skin sensations/redness (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (17) | 16 (16) — Feeling itchy or prickly sensations under the electrodes with/without skin redness

LIMITATIONS AND CAVEATS:
Enrollment disruptions due to COVID-19 pandemic resulted in a smaller size than planned (86%; n=62 across three groups out of n=72 planned) for primary outcome analysis and inadequate numbers (51%; n=37 across three groups out of n=72) for analyses of secondary MRI outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04152772/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04152772/ICF_002.pdf